CLINICAL TRIAL: NCT04974047
Title: A Phase 2, Multicenter, Open-label, 2-Cohort Study to Investigate the Efficacy and Safety of PET Guided Neoadjuvant Treatment With Tislelizumab (BGB-A317) Plus Chemotherapy/Chemoradiotherapy in Patients With Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Study of Tislelizumab in Participants With Resectable Esophageal Squamous Cell Carcinoma
Acronym: RATIONALE-213
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-213; CTR20211753 (Other: ChinaDrugTrials)
Record Dates: First submitted 2021-07-03; First posted 2021-07-23 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Resectable Esophageal Squamous Cell Carcinoma
Keywords: Tislelizumab; PET; Chemotherapy; Chemoradiotherapy
MeSH Terms: interventions — tislelizumab; Paclitaxel; Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Responder) (Experimental): Participants received induction therapy of one 21-day cycle with cisplatin and paclitaxel administered on Day 1. Following the induction phase, participants with a decrease in positron emission tomography (PET) Standardized Uptake Value (SUV)max ≥ 35% then received neoadjuvant therapy consisting of 200 mg tislelizumab on Day 1 of each 21-day cycle for 3 cycles and chemotherapy doublet (cisplatin + paclitaxel) for 2 cycles. After neoadjuvant treatment, participants were assessed for disease resectability and underwent surgical resection of the tumor approximately 4 to 6 weeks later.
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Cisplatin; Procedure: Surgical resection
- Cohort B (Non-responder) (Experimental): Participants received induction therapy of one 21-day cycle with cisplatin and paclitaxel administered on Day 1. Following the induction phase, participants with a decrease in PET SUVmax < 35% then received neoadjuvant therapy consisting of 200 mg tislelizumab on Day 1 of each 21-day cycle for 3 cycles and investigator-chosen chemotherapy doublet (paclitaxel + cisplatin or 5-fluorouracil + cisplatin) for 2 cycles plus concurrent radiotherapy. After neoadjuvant treatment, participants were assessed for disease resectability and underwent surgical resection of the tumor approximately 4 to 6 weeks later.
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Cisplatin; Drug: 5-fluorouracil; Radiation: Radiotherapy; Procedure: Surgical resection

INTERVENTIONS:
Drug: Tislelizumab — Administered intravenously on Day 1 of each 21-Day Cycle.
  Other Names: BGB-A317
Drug: Paclitaxel — 135 mg/m^2 administered intravenously on Day 1 of each 21-Day Cycle.
Drug: Cisplatin — 80 mg/m^2 administered intravenously on Day 1 of each 21-Day Cycle.
Drug: 5-fluorouracil — 1000 mg/m^2 administered intravenously over Day 1 through 4 of each 21-Day Cycle.
  Arms: Cohort B (Non-responder)
Radiation: Radiotherapy — 40 grays/20 fractions
  Arms: Cohort B (Non-responder)
Procedure: Surgical resection — Performed as indicated in the treatment arm.

SUMMARY:
The purpose of this study is to evaluate the pathological complete response (pCR) in participants receiving tislelizumab plus chemotherapy/chemoradiotherapy as neoadjuvant treatment.

DETAILED DESCRIPTION:
This study enrolled participants with esophageal squamous cell carcinoma who were eligible to have their tumor removed by surgery (also called surgical resection). The treatment phase of the study included the following:

* Induction therapy, in which participants received 1 cycle of chemotherapy;
* Neoadjuvant therapy (neoadjuvant refers to treatment that occurs before surgery, which can make the tumor easier to remove). In this study participants received neoadjuvant therapy based on their response to induction therapy. Response to induction therapy was assessed using the maximum standardized uptake value (SUVmax) measured using a Positron Emission Tomography (PET) scan. The SUV number refers to the level of brightness on the PET scan which reflects metabolic activity; increased metabolic activity can indicate cancerous growth.

  * Participants with a decrease in SUVmax of 35% or more after induction therapy received neoadjuvant treatment with tislelizumab plus chemotherapy.
  * Participants with a decrease in SUVmax less than 35% after induction therapy received neoadjuvant treatment with tislelizumab plus chemotherapy and radiotherapy.
* Surgery to remove the remaining tumor (resection) was to occur 4-6 weeks after completion of neoadjuvant treatment.

After surgery participants were followed until death, lost to follow-up, withdrawal of consent, or until the study was completed

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Histologically confirmed esophageal squamous cell carcinoma (ESCC).
* Stage cT1-2N+M0 and cT3NanyM0 (per The American Joint Committee on Cancer 8th Edition).
* Evaluation by the investigator to confirm eligibility for an R0 resection with curative intent.
* Adequate hematologic and organ function, defined by protocol-specified laboratory test results obtained within 14 days before first dose.

Key Exclusion Criteria:

* Ineligible for treatment with any of the chemotherapy doublets of protocol-specified chemotherapy.
* Any prior therapy for current ESCC, including investigational agents, chemotherapy, radiotherapy, targeted therapy agents, or prior therapy with an anti-programmed cell death protein-1, anti-programmed cell death protein ligand-1, anti-programmed cell death protein ligand-2, or any other antibody or drug specifically targeting T-Cell co-stimulation or checkpoint pathways.
* History of fistula due to primary tumor invasion.
* Participants with high risk of fistula or sign of perforation evaluated by investigator.
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days before first dose.

  * Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent) and topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption, and short course (≤ 7 days) of corticosteroid prescribed prophylactically or for the treatment of a non-autoimmune condition are permitted.
* Active autoimmune diseases or history of autoimmune diseases that may relapse.

  * Controlled Type I diabetes, hypothyroidism only requiring hormone replacement, controlled celiac disease, skin diseases (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* History of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases.
* With infections requiring systemic antibacterial, antifungal, or antiviral therapy, including tuberculosis infection.

  * Severe infections within 4 weeks before first dose, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
  * Receive therapeutic oral or intravenous antibiotics within 2 weeks before first dose.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tangdu Hospital, Xi'an, Shaanxi
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 study centers in China.
Period: Overall Study
Arm/Group | Cohort A (Responder) | Cohort B (Non-responder)
Started | 30 | 40
Surgical Resection Performed | 21 | 33
Completed | 0 | 0
Not Completed | 30 | 40
Not completed — Sponsor Ended Study | 20 | 22
Not completed — Death | 8 | 17
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Responder) | Cohort B (Non-responder) | Total
Number analyzed (Participants) | 30 | 40 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.16) | 63.1 (7.06) | 63.7 (7.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 24 | 38 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 40 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 40 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 30 | 40 | 70

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate
Description: The pCR rate was defined as the percentage of participants with absence of residual tumor in the resected primary tumor and all resected lymph nodes after completion of neoadjuvant treatment. pCR rates were assessed by a pathologist at each site.
Time Frame: pCR was determined from samples taken during surgery; surgery occurred 4-6 weeks after the last dose of chemotherapy, approximately Day 71-86
Population: The Efficacy Evaluable Analysis Set included all participants who received neoadjuvant treatment followed by surgery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Responder) | Cohort B (Non-responder)
Number analyzed (Participants) | 20 | 32
percentage of participants | 30.0 [11.9 to 54.3] | 34.4 [18.6 to 53.2]

2. Secondary Outcome: R0 Resection Rate
Description: Defined as the percentage of participants with R0 resection. R0 resection refers to a surgical procedure where the entire tumor is completely removed with no evidence of residual cancer tissue at the surgical margins.
Time Frame: Resection was planned to occur 4-6 weeks after the last dose of chemotherapy, approximately Day 71-86
Population: The Efficacy Evaluable Analysis Set included all participants who received neoadjuvant treatment followed by surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A (Responder) | Cohort B (Non-responder)
Number analyzed (Participants) | 20 | 32
percentage of participants | 95.0 | 90.6

3. Secondary Outcome: 1-year/3-year Disease-free Survival (DFS) Rate
Description: The DFS rate is defined as the percentage of participants free from disease events at 1 year and 3 years after the first date of no disease (R0 resection as surgery outcome). Disease events include local or distant recurrence or death due to any cause. The DFS rate was analyzed only for participants who underwent R0 resection. Disease-free rates were estimated using the Kaplan-Meier method with 95% confidence intervals estimated using the Greenwood formula.
Time Frame: 1 year and 3 years after surgery
Population: The Efficacy Evaluable Analysis Set with R0 resection included all participants who received neoadjuvant treatment followed by surgery with R0 resection. No participants were on follow-up for 3 years after surgery, so DFS rate at 3 years was not assessed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Responder) | Cohort B (Non-responder)
Number analyzed (Participants) | 19 | 29
percentage of participants
  1 Year | 79.0 [47.9 to 92.7] | 74.2 [53.3 to 86.8]
  3 Years: number analyzed (Participants) | 0 | 0

4. Secondary Outcome: 1-year/3-year Event-free Survival (EFS) Rate
Description: The EFS rate is defined as the percentage of participants free from EFS events at 1 year and 3 years after the first dose. The EFS events include progression of disease that precludes definitive surgery, local or distant recurrence, or death due to any cause. Event-free rates were estimated using the Kaplan-Meier method with 95% confidence intervals estimated using the Greenwood formula.
Time Frame: 1 year and 3 years after first dose date
Population: The Safety Analysis Set included all participants who received at least one dose of any component of study drugs.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Responder) | Cohort B (Non-responder)
Number analyzed (Participants) | 30 | 40
percentage of participants
  1 Year | 87.1 [64.3 to 95.8] | 67.8 [48.3 to 81.2]
  3 Years | 75.5 [49.8 to 89.3] | 59.9 [40.0 to 75.1]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is defined as the percentage of participants who have a complete response or partial response before surgery as assessed by the investigator per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) in all participants with measurable disease at baseline. Tumor response was assessed by computed tomography (CT) or magnetic resonance imaging (MRI) of the neck, chest, and abdomen.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: ORR was assessed prior to surgery, Day 71 to 86
Population: The Safety Analysis Set with Measurable Disease at Baseline included all participants who had measurable disease at baseline and received at least one dose of any component of study drugs.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (Responder) | Cohort B (Non-responder)
Number analyzed (Participants) | 21 | 33
percentage of participants | 71.4 [47.8 to 88.7] | 42.4 [25.5 to 60.8]

6. Secondary Outcome: Number Of Participants Experiencing Treatment-Emergent Adverse Events
Description: Immune-mediated AEs were reported until 90 days after the last dose of tislelizumab
Time Frame: From the first dose of study drug up to 30 days after last dose of any component of treatment or surgery or the initiation of subsequent anticancer therapy, whichever occurred first. Up to approximately 9 months.
Population: The Safety Analysis Set included all participants who received at least one dose of any component of study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Responder) | Cohort B (Non-responder)
Number analyzed (Participants) | 30 | 40
Participants | 30 | 39

ADVERSE EVENTS:
Time Frame: All-cause-mortality: From first dose until the end of study; maximum time on study follow-up was 37.3 months. AEs: From the first dose of study drug up to 30 days after the last treatment (any component of combination treatment or surgery, whichever is last) or the initiation of subsequent anticancer therapy, whichever occurred first. Immune-mediated AEs were reported until 90 days after the last dose of tislelizumab, up to approximately 9 months.
Arm/Group | Cohort A (Responder) | Cohort B (Non-responder)
All-Cause Mortality (participants affected / at risk) | 8/30 | 17/40
Serious Adverse Events (participants affected / at risk) | 8/30 | 12/40
Other Adverse Events (participants affected / at risk) | 30/30 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Responder) (N=30) | Cohort B (Non-responder) (N=40)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Anastomotic fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Responder) (N=30) | Cohort B (Non-responder) (N=40)
Anaemia (Blood and lymphatic system disorders) | 21 (30) | 32 (47)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 4 (4) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (18) | 14 (32)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 10 (16) | 16 (29)
Asthenia (General disorders) | 2 (4) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 7 (7)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 4 (5)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 8 (9)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 7 (7)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3)
Bile acids increased (Investigations) | 1 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 5 (7)
Blood creatinine increased (Investigations) | 3 (4) | 5 (6)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 2 (2)
Blood magnesium decreased (Investigations) | 1 (3) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 4 (6)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (8) | 9 (12)
Monocyte count decreased (Investigations) | 0 (0) | 3 (5)
Neutrophil count decreased (Investigations) | 19 (41) | 34 (75)
Neutrophil count increased (Investigations) | 1 (1) | 3 (3)
Platelet count decreased (Investigations) | 7 (10) | 12 (21)
Protein total decreased (Investigations) | 1 (1) | 8 (13)
Weight decreased (Investigations) | 3 (3) | 10 (10)
White blood cell count decreased (Investigations) | 19 (41) | 35 (85)
White blood cell count increased (Investigations) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (6) | 9 (9)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (6) | 10 (29)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (6)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (4) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (7) | 16 (22)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (11) | 11 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (7) | 5 (8)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (6)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 5 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Hypertension (Vascular disorders) | 2 (3) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT04974047/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT04974047/SAP_001.pdf